CLINICAL TRIAL: NCT03060499
Title: Post Thyroidectomy Myocardial Function
Acronym: TECH
Status: Withdrawn | Type: Observational
Why Stopped: Luck of interest
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Assistant Professor of Surgery, Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Other Study IDs: 584/13.10.2016
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Thyroid; Thyroidectomy; Myocardial Function
Keywords: Thyroidectomy; Myocardial Function; Thyroid gland; Heart
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol Synopsis

Protocol title: Post thyroidectomy myocardial function Purpose: Evaluation of the effects of total thyroidectomy on myocardial function Design: Prospective, single-center, cohort study Patient Population: Male or female subjects 18 years of age or older who are scheduled for total thyroidectomy No. of Subjects: 50 patients, estimated up to 12 months to enroll Duration of Treatment: Operation Duration of Follow-up: After discharge, the patients will be re-evaluated at three (3), six (6) and twelve (12) months in the outpatient clinic.

Endpoints: To evaluate the changes in the myocardial function after the removal of the thyroid gland.

DETAILED DESCRIPTION:
1.0 INTRODUCTION

It is commonly known that the thyroid hormones affect the function of the cardiovascular system. Several studies mention that these hormones influence the cardiac function and geometry directly and indirectly. Three potential mechanisms have been described, which are the direct cellular effect, the interaction with the sympathetic nervous system and changes in peripheral circulation.

A few studies have been already published , dealing with the correlation between thyroid hormones and heart function. Only one of them have proved a suppressed ventricular contractility after subtotal thyroidectomy for hyperthyroidism.

This clinical trial aims to compare the pre- and post-operative heart function after total thyroidectomy, using echocardiography. Outcomes will be assessed during patient hospitalization and at three, six and twelve months' follow-up appointments.

2.0 OBJECTIVES

To evaluate the effects of total thyroidectomy on the function of the cardiac muscle.

3.0 DESIGN AND STUDY POPULATION

The study is designed as a prospective, single-center, cohort study. Any patient that is scheduled for a total thyroidectomy will be offered participation in this study if they fulfill specific inclusion and exclusion criteria.

3.3 Duration of the study

The study will be conducted until at least 50 patients are treated. It is estimated that it will take up to 12 months to enroll the patients and an additional 12 months to complete follow-up assessments.

4.0 STUDY PROCEDURE

4.1 Pre-operative requirements

Procedures preformed such as routine hospital examinations, antibiotic prophylactic treatment, anticoagulant treatment and diet will be according to the standard management protocol and will be recorded for the study. The following pre-operative information will be recorded:

1. Demographic information including: name, age, gender, ethnicity
2. Height, weight, Body Mass Index (B.M.I.) and American Society of Anesthesiologists' (A.S.A.) physical status
3. Behavioral history (Smoking, alcohol or drug use)
4. Preoperative laboratory findings (Complete blood count, Ca2+, fT3, fT4, TSH, PTH, VitD)
5. Preoperative echocardiography
6. Diagnosis including clinical observation and previous imaging results
7. Medications
8. Current and past history of surgical and medical comorbidities

4.3 Pathology data

The following pathology data will be recorded for all patients:

1. Post-operative diagnosis including pathology report
2. Weight of the gland
3. Dimensions of the gland

4.4 Postoperative follow-up

Follow-up evaluation will be performed during hospitalization as well as on the 3rd, 6th and 12th month after discharge. The following information will be recorded:

1. Wound condition
2. Average Pain score for patient resting and moving/day
3. Postoperative laboratory findings (Complete blood count, Ca2+, fT3, fT4, TSH, PTH, VitD)
4. Postoperative echocardiography at three (3), six (6) and twelve (12) months.
5. Clinical signs of hypocalcemia (Chvostek and Trousseau)
6. Comments

5.0 COMPLICATIONS AND ADVERSE EVENTS

The investigators are required to notify the coordinators of any serious adverse events. The coordinators are also required to notify the Ethics Committee according to local regulations and requirements.

Serious Adverse Events include:

1. Death regardless of cause
2. Any-life-threatening event
3. Any hospitalization or prolongation of existing hospitalization
4. Any event that results in persistent or significant disability or incapacity to the patient.

6.0 STATISTICAL ANALYSIS

The objective of this study is to evaluate the effects of total thyroidectomy on the myocardial function.

Statistical analysis includes description of the pre- and post-operative outcomes, and indication of patient characteristics associated with these outcomes.

Since the study does not have pre-specified hypotheses all statistical analyses are exploratory and interpretation of results should be within this context.

7.0 DATA MONITORING PLAN

The coordinators will monitor all data. Furthermore, the coordinators will review the progress of the clinical trial including safety data and ensure that it is conducted, recorded and reported in accordance with the protocol, good clinical practice and the applicable regulatory requirements.

8.0 DATA CONFIDENTIALITY

Each patient will be identified by his/her initials and a unique patient identification number. Source data will be stored with source documents. Only personnel responsible for collecting data and transcribing it into the case report forms will have access to the data. Records will be protected.

9.0 FUNDING

No funding for the execution of the present protocol is considered necessary. The investigators are willing to execute the present study without any additional reimbursement.

10.0 ETHICS

Prior to the onset of the study, institution review board (IRB) approval should have been obtained. Any changes in the study protocol, informed consent forms, or investigator must be re-approved by the IRB. All patients enrolled in the study will provide their consent prior to entering the study. Informed consent forms shall be signed and dated by the patient. The investigator will retain the forms as part of the study records.

This study will be executed in accordance with the Declaration of Helsinki, in agreement with the guidelines for conducting a clinical investigation and the principles of ICH GCP outlined in the E6 document. By signing the present protocol, participants in the study commit themselves to carry it out with respect to local legal requirements.

11.0 INFORMED CONSENT

All eligible patients should have the capacity to provide an written informed consent.

The above described inclusion and exclusion criteria were designed to ensure the entry of the appropriate population of patients to this study and will be approved by the local IRB. Screening for these criteria will be conducted by the coordinator.

Eligible patients will be educated about the research proposal by a study investigator. To determine whether the patient has understood the issues, they will be asked to describe what the research entails and whether they have any questions. All questions will be addressed prior to enrollment. The patient can decline participation in the study at any time.

A written informed consent form will be generated. For each patient, a case report form (CRF) will be completed, providing general medical information and history.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years old
* Patient scheduled for a non-emergency operation
* Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures
* No previous cardiologic history
* Normal PTH values (no transient hypoparathyroidism)

Exclusion Criteria:

* Patient is underage ( under 18 years old)
* Patient had a previous operation at the thyroid or parathyroids
* Patient inability to participate in follow-up appointments
* Patient is participating in another clinical trial which may affect this study's outcomes
* Patient with TSH values outside the range of normal values
* Pathologic Ca2+ , Vit D, P, PTH, pre- and post-operative values
* Diabetes Mellitus, Hypertension, History of any heart, lung or systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is designed as a prospective, single-center, cohort study. Any patient that is scheduled for a total thyroidectomy in 1st Propedeutic Department of Surgery (AHEPA University General Hospital) will be offered participation in this study if they fulfill the following requirements.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-10-13 (Estimated); Study Completion 2018-10-13 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic Assessment of Changes in Myocardial Function at 3, 6 and 12 months after Thyroidectomy | They will be assessed at 3, 6 and 12 months after thyroidectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Pliakos, Academic Fellow, Principal Investigator — 1st Propedeutic Department of Surgery, AHEPA University General Hospital, Aristotle University of Thessaloniki; Antonios Michalopoulos, Professor, Principal Investigator — 1st Propedeutic Department of Surgery, AHEPA University General Hospital, Aristotle University of Thessaloniki; Georgios Efthimiadis, Assistant Professor, Principal Investigator — 1st Cardiology Unit, AHEPA University General Hospital, Aristotle University of Thessaloniki; Haralambos Karvounis, Professor, Principal Investigator — 1st Cardiology Unit, AHEPA University General Hospital, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University General Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bengel FM, Nekolla SG, Ibrahim T, Weniger C, Ziegler SI, Schwaiger M. Effect of thyroid hormones on cardiac function, geometry, and oxidative metabolism assessed noninvasively by positron emission tomography and magnetic resonance imaging. J Clin Endocrinol Metab. 2000 May;85(5):1822-7. doi: 10.1210/jcem.85.5.6520. PMID 10843159
- [Background] Polikar R, Burger AG, Scherrer U, Nicod P. The thyroid and the heart. Circulation. 1993 May;87(5):1435-41. doi: 10.1161/01.cir.87.5.1435. PMID 8490997